CLINICAL TRIAL: NCT07200986
Title: A Phase 1, Randomized, Double-blind, Two-arm, Parallel-Group, Single-dose Study to Compare Pharmacokinetics and Safety of CT-P52 and US-licensed Taltz in Healthy Subjects
Brief Title: Study to Compare Pharmacokinetics and Safety of CT-P52 and US-licensed Taltz in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P52 1.1
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — ixekizumab

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, two-arm, parallel-group, single-dose study designed
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P52 (Experimental): 80 mg (single dose), subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: Ixekizumab
- United States (US)-licensed Taltz (Active Comparator): 80 mg (single dose), subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: Ixekizumab

INTERVENTIONS:
Biological: Ixekizumab — 80 mg (single dose), SC injection via PFS

SUMMARY:
This study is designed to demonstrate PK similarity of the proposed biosimilar test product CT-P52 and the reference product, US-licensed Taltz.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 19 to 55 years, both inclusive.
* Subject with a body weight of ≥60 and ≤90 kg for male and ≥50 and ≤90 kg for female, and a BMI between 18.0 and 29.9 kg/m2 (both inclusive) when rounded to the nearest tenth.
* Subject is able to understand and to comply with protocol requirements, instructions, and restrictions.

Exclusion Criteria:

* A medical history and/or condition that is considered significant
* Clinically significant allergic reactions, hypersensitivity
* History or current infection of human immunodeficiency virus, hepatitis B virus, hepatitis C virus or syphilis
* Active or latent Tuberculosis
* Previous monoclonal antibody or fusion protein treatment, or current use of any biologics
* Plans to donate whole blood or blood components during the study
* Male subject who is planning to have child or donate sperms within 10 weeks after the study drug administration. Female subject who is currently pregnant or lactating, or planning to be pregnant or to breastfeed within 10 weeks after the administration of the study drug
* Reasonable evidence or history of drug/alcohol/smoking abuse
* Presence of tattoos, sunburn, or other skin disturbances on the injection site
* Vulnerable subject

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
AUC0-inf | Day 85
  Pharmacokinetic (PK) similarity demonstration in terms of area under the concentration-time curve (AUC) from time zero to infinity (AUC0-inf)
Cmax | Day 85
  PK similarity demonstration in terms of maximum serum concentration

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan, Busanjin-gu
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided